CLINICAL TRIAL: NCT05059483
Title: Psychometric Evaluation of the Spanish Version of the Physiotherapy Critical Thinking in Clinical Practice Questionnaire: Multicenter Study
Brief Title: Physiotherapy Critical Thinking in Clinical Practice Questionnaire
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PT-CT-4 Practice
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-01

CONDITIONS: Critical Thinking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
A greater need for user-centered care and an evidence-based clinical practice are factors that emphasize critical thinking as a professional competence. Furthermore, critical thinking is an essential competence that allows clinical reasoning, problem solving and decision-making in the critical clinical practice of all specializations in Physiotherapy. However, no instrument has been found that specifically assesses the critical thinking of physiotherapists in their clinical practice.

DETAILED DESCRIPTION:
Multicenter, descriptive, cross-sectional and correlational study in two phases. Phase 1: adaptation of the N-CT-4P to the population of physiotherapists; Phase 2: analysis of the psychometric properties of the new instrument and levels of critical thinking through a cross-sectional study. Sociodemographic and professional variables and variables referring to the measurement of critical thinking (total score of the questionnaire and of each of its dimensions) will be collected. Its psychometric properties, internal consistency, repeatability analysis, discriminant validity and construct validity will be analyzed through confirmatory factor analysis and a multiple regression analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Be a Graduate, Diploma or Bachelor of Physiotherapy
* Have an employment contract, as a care physiotherapist at the time of answering the questionnaire.

Exclusion Criteria:

* Have a contractual continuity of less than 15 days.

Ages: 18 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Health centers
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
To validate in the physiotherapist population the instrument Nursing Critical Thinking in Clinical Practice Questionnaire (N-CT-4 Practice) in its version Physiotherapy Critical Thinking in Clinical Practice Questionnaire (PT-CT-4 Practice). | The questionnaire will be self-administered and the estimated response time is less than 15 minutes.
  Assessment of metric properties

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Hernández-Méndez, MSc, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute; Esperanza Zuriguel-Pérez, PhD, Study Chair — Hospital Universitari Vall d'Hebron Research Institute
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Hernandez-Mendez B, Gines-Puertas A, Jerez-Roig J, Marti-Romeu JD, Camara-Menoyo D, Cuartero-Archs J, Piqueras-Cespedes M, Llaberia-Marcual M, Zuriguel-Perez E. Psychometric evaluation of the Spanish version of the physiotherapy critical thinking in clinical practice questionnaire. Clin Rehabil. 2025 Oct;39(10):1355-1365. doi: 10.1177/02692155251362999. Epub 2025 Jul 31. PMID 40739927